CLINICAL TRIAL: NCT01945788
Title: Comparación de la Eficacia y Seguridad clínicas de Osteofortil Respecto de Forteo
Brief Title: Clinical Comparison of Efficacy and Safety of Two Teriparatide Formulations: Osteofortil and Forteo
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bio Sidus SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1301
Record Dates: First submitted 2013-09-11; First posted 2013-09-19 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2013-09

CONDITIONS: Postmenopausal Osteoporosis With Pathological Fracture
MeSH Terms: interventions — Teriparatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Teriparatide Forteo (Active Comparator): 20 micrograms/day plus calcium and vitamin D
  Interventions: Drug: Teriparatide (rDNA origin)
- Teriparatide Osteofortil (Experimental): 20 micrograms/day plus calcium and vitamin D
  Interventions: Drug: Teriparatide (rDNA origin)

INTERVENTIONS:
Drug: Teriparatide (rDNA origin)

SUMMARY:
The primary objective of this study is to compare efficacy and safety of two formulations of teriparatide 20 mcg/day plus calcium and vitamin D in postmenopausal women with osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

I. Female.

II. Age greater than or equal to 50 and less than 81 years.

III. Last menstrual period at least one year prior to signing the informed consent.

IV. Osteoporosis. Defined by the presence of:

BMD by DEXA with a T-score of -2.5 or lower on lumbar spine or T-score at the lumbar spine, femoral neck or total hip -2.0 or below, together with one or more vertebral fractures documented by lateral spine radiographs.

V. Have signed the informed consent

-

Exclusion Criteria:

I Bone alkaline phosphatase in the blood above the normal limit without any explanation.

II. Liver disease (AST or ALT> 2 x ULN). III. Renal disease (serum creatinine> 2.0 mg / dl) and / or creatinine clearance <30 ml / min IV. Hypercalcemia ([Ca]> 10.5 mg / dL). Patients with elevated PTH in the presence of albumin-corrected calcium within normal values can be re-evaluated.

V. Elevated blood PTH ([PTH]> 65 pg / ml) Patients with elevated PTH in the presence of albumin-corrected calcium within normal values can be re-evaluated.

VI. • Deficiency of vitamin D (25-OH vitamin D <16 ng / ml) or excess vitamin D (above 80 ng / ml blood). Patients who did not meet the inclusion criteria for vitamin D may receive a supplement (vitamin D) and be re-evaluated.

VII. • Anemia (hematocrit <32%).

VIII. • History of cancer (except basal cell carcinoma) or radiotherapy.

IX. Severe cardiopulmonary disease, including coronary heart disease: unstable angina, heart failure class III or IV or any other condition that the investigator believes may prevent participation safely and complete the protocol procedures.

X. Major psychiatric disease that in the opinion of the investigator, would prevent to give properinformed consent or complete the study procedures.

XI. Excessive alcohol or substance abuse that in the opinion of the investigator prevents giving informed consent or complete proper protocol procedures.

XII. Congenital or acquired bone disease, other than osteoporosis (including osteomalacia, hyperparathyroidism or Paget's disease)

XIII. Regarding the history of ingestion of oral bisphosphonates: After assessment of adequate adherence (compliance greater than 75%), if the patient received six months of treatment, she should have a bisphosphonate-free period of six months. If she took more than six months, the bisphosphonate-free period must be 12 months.

XIV. Current or within the last 3 months before study entry estrogen use, selective estrogen receptor modulators use or calcitonin use in therapeutic doses.

XV. Current use of systemic corticosteroids (oral or parenteral) for more than 14 days in the last 6 months. Vaginal estrogen and isoflavones are permitted .

XVI.Current or previous use of teriparatide, other PTH analogues as patches or injectables, strontium, fluorine or any intravenous bisphosphonate therapeutic dose, XVII. Known hypersensitivity to pharmaceuticals derived from bacterial cells. XVIII. Hypersensitivity to teriparatide or to any of its excipients. XIX.Nephrolithiasis or urolithiasis in activity, according to the investigator opinion in the 5 years prior to randomization.

XX.Inflammatory bowel disease, malabsorption syndrome or any sign of intestinal calcium malabsorption

XXI. Treatment with androgens or anabolic steroids in the 6 months prior to randomization.

XXII. Any medical condition that in the investigator opinion would contraindicate treatment with an investigational drug.

XXIII. Treatment with coumarin and indandione derivatives in the 3 months prior to randomization or treatment with heparins (at doses> 10,000 U / day) for more than 30 days in the 6 months prior to randomization.

XXIV.Treatment with any other drug known to affect bone metabolism, in therapeutic doses,in the 6 months prior to randomization.

XXV.Treatment with an investigational drug during the month prior to randomization. -

Ages: 50 Years to 81 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-10 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Bone mineral Density at 6 months. | Basal, Six months and One Year

SECONDARY OUTCOMES:
Change from baseline in P1NP, Osteocalcin, C-terminal cross-linked telopeptide of type I collagen levels at 3 and 6 months | Basal, 3, 6 and 12 months

OTHER OUTCOMES:
Change from baseline on bone mineral density asessed by High-resolution peripheral quantitative computed tomography (HR-pQCT) at 6 months | Basal, six months and one year.
Number of patients with elevated serum calcium | Basal, 1, 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Investigaciones Metabolicas, Buenos Aires, Buenos Aires F.D., Argentina